CLINICAL TRIAL: NCT03540368
Title: The Role of Tranexamic Acid for the Treatment of Gastrointestinal Bleeding: A Randomized Double-blind Controlled Trial
Brief Title: Tranexamic Acid for The Treatment of Gastrointestinal Bleeding
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: increased number of patients death
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ari Fahrial Syam, Medical Doctor, Gastroenterology Hepatology Consultant, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-04-0393
Record Dates: First submitted 2018-05-15; First posted 2018-05-30 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Gastrointestinal Bleeding
Keywords: Gastrointestinal bleeding; Tranexamic acid; Clinical trial
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Masking Description: All patients will receive standard treatment equally
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid injection (Experimental): Group with tranexamic acid injection
  Interventions: Drug: Tranexamic acid injection
- Placebo (Placebo Comparator): Group with Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tranexamic acid injection — Administering tranexamic acid loading dose 1 gram in 100 cc sodium chloride 0,9%, followed by maintenance dose 3 grams in infusion for 24 hours.
  Arms: Tranexamic acid injection
Other: Placebo — Administering placebo or sodium chloride 0,9% intravenously
  Arms: Placebo

SUMMARY:
Studies showed that in cases of gastrointestinal bleeding, injection tranexamic acid decreasing the risk of death and the need of surgical intervention. However, the quality of most clinical trials were not good and the results were not significant. Injection tranexamic acid does not become one of the treatment option in the international guidelines nor in national consensus, so the effectiveness and the safety of its use in the treatment of gastrointestinal bleeding remains unclear and not routinely used.

In Indonesia, injection tranexamic acid in gastrointestinal bleeding is limitedly used and recorded. Therefore, a clinical trial study of injection tranexamic acid is required to assess the effectiveness and the safety in the treatment of gastrointestinal bleeding.

DETAILED DESCRIPTION:
This study is a randomized double-blind controlled trial study. Interventions were given in the form of tranexamic acid injection compared to placebo in patients with acute upper and lower gastrointestinal bleeding. Tranexamic acid were administered intravenously 1 gram loading dose, followed by 3 grams maintenance dose in infusion for 24 hours. Other routine and standardized drugs for gastrointestinal bleeding will still be given. Statistical analysis will use: Chi square test or Kolmogorov-Smirnov with alternative Fisher test for categorical dependent-variable; Independent T-Test with alternative Mann-Whitney test for two-group numerical dependent-variable; and one-way ANOVA with alternative Kruskal-Wallis for more than two-groups numerical dependent-variable.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Patients with acute lower and upper gastrointestinal bleeding (assessed clinically)
* Patients agreed to participate in the study and signed the informed consent

Exclusion Criteria:

* Allergy with tranexamic acid
* Patients considered by the clinician can not be randomized to participate in the study
* Patients with chronic kidney disease stage III - V

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2018-07-04 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Re-bleeding | 30 days after randomisation
  Total incidence number of re-bleeding

SECONDARY OUTCOMES:
Number of death | 30 days after randomisation
  Total number patients who die
Need for blood transfusion | 30 days after randomisation
  Total number of patients with blood transfusion
Length of stay in intensive care unit | 30 days after randomisation
  Average time of stay each participants in intensive care unit
Need for endoscopic hemostasis | 30 days after randomisation
  Total number of patients with endoscopic hemostasis
Quality of life (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health) | 30 days after randomisation
  Short Form-36 Questionnaire includes one scale for each of eight measured health domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. All health domain scales are scored using norm-based scores ranging 0 to 100 with higher scores indicate better health
Level of anxiety | 30 days after randomisation
  Hamilton Anxiety Rating Scale; Each item is scored of 0 (not present) to 4 (severe), with total score range of 0-56, where <14 indicates no anxiety, 14-20 mild anxiety, 21-27 moderate anxiety, 28-41 severe anxiety and 42-56 very severe anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Ari F Syam, Dr, MD, Principal Investigator — Gastroenterology Division, Internal Medicine Department RSCM/UI
Locations (1):
- Cipto Mangunkusumo National Central General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bennett C, Klingenberg SL, Langholz E, Gluud LL. Tranexamic acid for upper gastrointestinal bleeding. Cochrane Database Syst Rev. 2014 Nov 21;2014(11):CD006640. doi: 10.1002/14651858.CD006640.pub3. PMID 25414987

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT03540368/Prot_SAP_001.pdf